CLINICAL TRIAL: NCT06734429
Title: Management of Patients Who Had an Artificial Urethral Sphincter by Laparotomy in Childhood
Brief Title: Urinary Artificial Sphincter in Children
Acronym: SUAPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Destinval Christelle, Dr., University Hospital, Clermont-Ferrand
Other Study IDs: M24DC1105
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Neurogenic Bladder Disorder; Bladder Dysfunction; Spina Bifida; Urinary Incontinence Due to Urethral Sphincter Incompetence; Child, Only
Keywords: Urinary Artificial Sphincter; Neurogenic Bladder; Child; Outcomes; Retrospective Study
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Dysraphism | interventions — Urinary Sphincter, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Urinary Artificial Sphincter (UAS) in Children: Patients aged under 18 years old with UAS
  Interventions: Other: Urinary Artificial Sphincter

INTERVENTIONS:
Other: Urinary Artificial Sphincter — Urinary Artificial Sphincter is a device used for patients with urethral sphincter incompetence

SUMMARY:
Retrospective monocentric study of the outcomes of patients with neurogenic bladder who had a urinary artificial sphincter before the age of 18 years old. Hypothesis: what was the impact of the urinary artificial sphincter on the global management of the patient?

DETAILED DESCRIPTION:
The management of patients with neurogenic bladder is complex. Several patients have been operated multiple times. Surgical procedures such as Mitrofanoff's, bladder neck surgery, bladder augmentation, and urinary artificial sphincter are common. The investigators wanted to analyze the participants' data, which led to the indication of a urinary artificial sphincter and its outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were younger than 18 years old when they had an urinary artificial sphincter

Exclusion Criteria:

* Patients who were 18 years old or older when they had an urinary artificial sphincter

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients younger than 18 years old who have neurogenic bladders
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with urinary sphincter incomptetence | Before surgery
  Participants with urinary incontinence caused by urinary sphincter incomptetence
Impact of urinary artificial sphincter on the participants' incontinence | Through study completion, an average of 2 years
  Three outcomes are possible: the participant is continent (with or without a few leaks), the participant is continent with catheterization, the patient is incontinent.

SECONDARY OUTCOMES:
Impact of bladder augmentation on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of bladder augmentation in participants with urinary artificial sphincter. Three outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.
Impact of Mitrofanoff procedure on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of Mitrofanoff procedure in participants with urinary artificial sphincter. Three outcomes are possible: the participant is continent, the participant is continent with catheterization, or the patient is incontinent.
Impact of bladder neck surgery on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of bladder neck surgery in participants with urinary artificial sphincter. hree outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.
Last follow-up | Through study completion, an average of 2 years]
  Follow-up represents the time between the surgery and postoperative consultation dates in days, months, or years.
  Generally, there are a-month-follow-up, a three month-follow-up, a six month-follow-up, and a year-follow-up. The surgeon can see the patient if there is any problem between these consultations. After a year of follow-up, it is up to the surgeon to decide if the patient needs to be seen yearly or not. The last follow-up date is crucial because it indicates how the patient is and if other follow-up dates need to be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization the investigators won't share individual participant data

REFERENCES:
- [Background] Delgado-Miguel C, Munoz-Serrano A, Amesty V, Rivas S, Lobato R, Martinez-Urrutia MJ, Lopez-Pereira P. Artificial urinary sphincter in congenital neuropathic bladder: Very long-term outcomes. Int J Urol. 2022 Jul;29(7):692-697. doi: 10.1111/iju.14874. Epub 2022 Mar 26. PMID 35340070